CLINICAL TRIAL: NCT03405974
Title: Aspirin (Acetylsalicylic Acid) in the Prevention of Collapse of the Femoral Head in Early-stage Non-traumatic Osteonecrosis: a Two-year Multicenter, Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Aspirin in the Prevention of Collapse in Osteonecrosis of the Hip
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Chantal Seguin, Hematologist-oncologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONFH-ASA2016
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Osteonecrosis of Femoral Head; Osteonecrosis; Aseptic, Idiopathic
Keywords: Osteonecrosis; Aspirin
MeSH Terms: conditions — Femur Head Necrosis; Osteonecrosis; Infertility | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective, randomized, double-blind, placebo-controlled trial that aims to test the efficacy of the proposed medical intervention (ASA). The design is intended to be parallel group where a total of 114 patients will be randomized in a 1:1 ratio to the treatment (ASA) and the control (Placebo) arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of ASA and Placebo treatments will not be known to investigators, research staff, or patients. Access to the randomization code will be strictly controlled in order to ensure double-blind administration of study treatments. Packaging and labeling of ASA and Placebo treatments will be identical to maintain the blind.
  All of the study drug profiles will be prepared in order to be identical in appearance to preserve the study blinding. The investigator and the subject, as well as all staff involved in the conduct or management of the study will be blinded to which treatment is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Aspirin 100 mg
  1 tablet/ day for 2 years
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo
  1 tablet/ day for 2 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin (acetylsalicylic acid)
  Other Names: acetylsalicylic acid
  Arms: Aspirin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if prolonged administration of low-dose aspirin will prevent the progression of early-stage osteonecrosis of the femoral head and may even reduce the extent of involvement of the femoral head by the necrotic process The design is intended to be parallel group where a total of 114 patients will be randomized in a 1:1 ratio to the treatment (ASA) and the control (Placebo) arms.

DETAILED DESCRIPTION:
1. TRIAL OBJECTIVES The primary objective of this study is to evaluate the radiologic progression of ONFH on either radiographs or MRI. A successful outcome is defined as no difference in ONFH staging according to the Ficat & Arlet or Steinberg classifications at last patient follow-up compared to initial radiological staging. This translates into lack of progression over the course of the study while the natural evolution is progression over time.

   The secondary objective is to evaluate the percentage of involvement of the femoral head on radiographs and/or MRI which measures the extent of the disease. We expect that the extent of the disease will be reduced at 2 years.
2. STUDY DESIGN AND DURATION This study is a multicenter, prospective, randomized, double-blind, placebo-controlled trial that aims to test the efficacy of the proposed medical intervention (ASA). The design is intended to be parallel group where a total of 114 patients will be randomized in a 1:1 ratio to the treatment (ASA) and the control (Placebo) arms.

All patients presenting to the osteonecrosis clinic of one of the participating centres will be first evaluated by an orthopedic surgeon to confirm the diagnosis of early ONFH on at least one hip. Selected patients will be screened for eligibility according to specific inclusion and exclusion criteria.

Eligible patients who accept to participate in this study will be randomized to either a control arm (placebo) or a treatment arm (Aspirin). Recruited patient will take their assigned treatment daily at breakfast from enrolment and for a minimum of two years They will be followed over a period of 2 years. Evaluations will be taken at baseline and every 6 months (5 visits in total).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old
2. Patients with early osteonecrosis of the hip as defined above
3. Diagnosis confirmed within 3 months of the screening visit
4. Patients accept to take the study medication

Exclusion Criteria:

1. A history of hip trauma or surgery affecting the hip involved with early stage osteonecrosis as per criteria above
2. Concurrent use of anticoagulants
3. Concurrent use of bisphosphonates
4. Concurrent use of Aspirin for any reason
5. Patients with recent active severe peptic ulcer disease that are not on PPI.
6. Patients with advanced osteonecrosis of the hip with signs of collapse or end-stage joint arthritis of the hip that are immediately referred for surgical consultation for THA
7. Patients who are hypersensitive to ASA, salicylates, or non-steroidal anti-inflammatory drugs
8. Hepatic impairment (Bilirubin total, AST, ALT > 2-3x upper limit of normal), renal failure (creatinine level above normal with glomerular filtration rate < 45 ml/minute), or congestive heart failure
9. Platelets number should be more than 100,000 ( > 100 x 109 /L)
10. Pregnancy. If the patient is not sure whether she may be pregnant or not, a screening for pregnancy should be done.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of radiologic progression of osteonecrosis | 6 months
  The primary endpoint is to evaluate the radiologic progression of ONFH by measuring the difference in ONFH staging according to the Ficat & Arlet or Steinberg classifications at last patient follow-up compared to initial radiological staging.

SECONDARY OUTCOMES:
Measure the percentage involvement of the femoral head on MRI. | 6 months
  The secondary endpoint is to measure evolving extent of involvement of the femoral head on radiographs and/or MRI that measures the extent of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Séguin, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albers A, Carli A, Routy B, Harvey EJ, Seguin C. Treatment with acetylsalicylic acid prevents short to mid-term radiographic progression of nontraumatic osteonecrosis of the femoral head: a pilot study. Can J Surg. 2015 Jun;58(3):198-205. doi: 10.1503/cjs.016814. PMID 26011853